CLINICAL TRIAL: NCT06224868
Title: Comparison of the Effects of Different PEEP Values With USG on Optic Nerve Sheath Diameter (ONSD), Diaphragmatic Thickness ,and Lung Score in Laparoscopic Surgery Patients
Brief Title: Comparison of the Effects of Different PEEP Values With USG on Optic Nerve Sheath Diameter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Begüm Nemika Gökdemir, Research Assistant, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: KA 23/230
Record Dates: First submitted 2024-01-02; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Cholecystitis
Keywords: laparoscopic surgery; pneumoperitoneum; optic nerve sheath diameter
MeSH Terms: conditions — Cholecystitis; Pneumoperitoneum | interventions — Insufflation

STUDY DESIGN:
Intervention Model Description: Group 1: PEEP 0 Group 2: PEEP 5 Group 3: PEEP 10
Who Masked: Participant, Investigator
Masking Description: The anesthesiologist will not tell the radiologist making ultrasonography (USG) measurements which PEEP she set on the mechanical ventilator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PEEP 0 (Active Comparator): After the patient is intubated, PEEP 0 will be set on the mechanical ventilator.
  Interventions: Other: insufflation; Other: desufflation
- PEEP 5 (Active Comparator): After the patient is intubated, PEEP 5 will be set on the mechanical ventilator.
  Interventions: Other: insufflation; Other: desufflation
- PEEP 10 (Active Comparator): After the patient is intubated, PEEP 10 will be set on the mechanical ventilator.
  Interventions: Other: insufflation; Other: desufflation

INTERVENTIONS:
Other: insufflation — Laparoscopic surgery begins with intraabdominal placement of the insufflation needle or trochar, followed by carbon dioxide (CO2) insufflation of the abdominal cavity to an intraabdominal pressure (IAP) of 12 to 15 mm Hg (Normal values are 5-7 mmHg) it is aimed to monitor optic sheat nerve diameter and lung ultrasound score changes with different intraabdominal pressures.
Other: desufflation — Laparoscopic surgery begins with intraabdominal placement of the insufflation needle or trochar, followed by carbon dioxide (CO2) insufflation of the abdominal cavity to an intraabdominal pressure (IAP) of 12 to 15 mm Hg. When the surgery is completed, the trochars are removed and intra-abdominal pressure is returned to normal which is 5-7 mmHg.

SUMMARY:
Laparoscopic surgeries are now more popular because of the advantages such as shorter hospital stay, minimal scar. In order to perform laparoscopic surgery, pneumoperitoneum should be initiated. The optic nerve sheath is an extension of the dura mater and the subarachnoid space is continuous with the intracranial subarachnoid space. Therefore, non-invasive monitoring of the increase in intracranial pressure (ICP) can be achieved by measuring the optic nerve and sheath diameter with ultrasound. Since ONSD measurement with ultrasound is an easily applicable technique, it is useful in monitoring intracranial pressure changes based on the optic nerve diameter during intraoperative changes

DETAILED DESCRIPTION:
Laparoscopic surgeries are now becoming increasingly common compared to traditional laparotomies, as they have advantages such as more minimal scarring, shorter hospital stay, fewer complications, and early mobilization. In these surgeries, pneumoperitoneum provided with carbon dioxide (CO2) has many effects on the cardiovascular, pulmonary, renal, metabolic and cerebral systems. Pulmonary compliance and functional residual capacity decrease due to pnemoperitoneum, ventilation/perfusion mismatch occurs, and as a result, hypoxemia may occur. A minimum of 4-6 cm H20 positive end-expiratory pressure (PEEP) should be applied to all intubated patients under general anesthesia to reduce postoperative pulmonary complications (especially atelectasis) and prevent ventilation/perfusion mismatch and hypoxemia. The optic nerve sheath is an extension of the dura mater and the subarachnoid space is continuous with the intracranial subarachnoid space. Therefore, non-invasive monitoring of the increase in intracranial pressure (ICP) can be achieved by measuring the optic nerve and sheath diameter with ultrasound. When ICP is > 20 mm Hg, measuring the optic nerve sheath diameter (ONSD) between 5.2 and 5.9 mm has a sensitivity of 74-95% and a specificity of 74-100%. Since ONSD measurement with ultrasound is an easily applicable technique, it is useful in monitoring intracranial pressure changes based on the optic nerve diameter during intraoperative changes (trendelenburg/reverse trendelenburg position, pneumoperitoneum , PEEP in mechanical ventilation).

ELIGIBILITY:
Inclusion Criteria:

* 18- 65 aged all female and male volunteers

Exclusion Criteria:

* acute or chronic eye diseases,
* uncontrolled hypertension,
* asthma
* known lung disease,
* body mass index (BMI) over 35 kg/m2,
* devices using bulbs with known intracranial charging,
* who refuse to participate in care

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
comparison of diameter of optic nerve sheath with ultrasonography (USG) for different PEEP values | Intraoperatively
  comparison of diameter of optic nerve sheath (ONSD) for different PEEP values with ultrasonography (Group 1: 0 cmH2O, Group 2: 5 cmH2O, Group 3: PEEP 10 cmH2O)
comparison of diaphragmatic thickness with USG for different PEEP values | Intraoperatively
  comparison of diaphragmatic thickness with USG for different PEEP values (Group 1: 0 cmH2O, Group 2: 5 cmH2O, Group 3: PEEP 10 cmH2O)
comparison of lung ultrasound scores (LUS) via USG for different PEEP values | Intraoperatively
  comparison of lung scores with USG for different PEEP values (Group 1: 0 cmH2O, Group 2: 5 cmH2O, Group 3: PEEP 10 cmH2O). This measurement calculated by
  LUS assigns 0 points to A lines or < 2 separate B lines plus regular sliding; 1 point with lines B ≥ 3 or spaced focal points plus regular sliding; 2 points with coalescing B lines, and 3 points to pulmonary consolidations with a score ranging from 0 (normal lungs) to 36 (worst case scenario)

SECONDARY OUTCOMES:
comparison of diameter of optic nerve sheath via USG with different intraabdominal pressures. | Intraoperatively
  comparison of diameter of optic nerve sheath via USG with different intraabdominal pressures. ( insufflation and desufflation) Laparoscopic surgery involves insufflation of a gas (usually carbon dioxide) into the peritoneal cavity producing a pneumoperitoneum.
  Normal intraabdominal pressure is 5-7 mmHg. Pneumoperitoneum is achieved by insufflation of the abdominal cavity to an intraabdominal pressure (IAP) of 12 to 15 mm Hg.
comparison of diaphragmatic thickness with USG with different intraabdominal pressures. | Intraoperatively
  comparison of diaphragmatic thickness with USG in different intraabdominal pressures ( insufflation and desufflation) Laparoscopic surgery involves insufflation of a gas (usually carbon dioxide) into the peritoneal cavity producing a pneumoperitoneum.
comparison of lung ultrasound scores (LUS) via USG with different intraabdominal pressures. | Intraoperatively
  comparison of lung ultrasound scores (LUS) via USG with different intraabdominal pressures. ( insufflation and desufflation)

IPD SHARING:
Plan to Share IPD: No